CLINICAL TRIAL: NCT06151990
Title: Assessment of Lipid Profile in Juvenile Systemic Lupus Erythematosus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Abdelnasser Mahmoud, principal investigator, Assiut University
Other Study IDs: lipid profile in JSLE
Record Dates: First submitted 2023-11-13; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-09

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- newly diagnosed juvenile systemic lupus erythematosus
  Interventions: Other: lipid profile
- old cases of juvenile systemic lupus in activity
  Interventions: Other: lipid profile
- old cases of juvenile systemic lupus not in activity(controlled)
  Interventions: Other: lipid profile

INTERVENTIONS:
Other: lipid profile — Measurements for CHOL,TG,LDL-C and HDL-C obtained following an overnight fasting

SUMMARY:
. To determine pattern and frequency of dyslipoproteinemia in patients with newly diagnosed juvenile SLE and to assess effect of disease activity on lipid profile of patients with juvenile SLE.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic autoimmune disease characterized by multisystem inflammation and the presence of circulating autoantibodies against self-antigens leading to inflammatory damage of many target organs including the skin, joints, kidneys, blood cells, blood vessels, and the central nervous system.Premature atherosclerosis has been recognized as an important issue for patients with SLE since the mid-1970s. Among the traditional risk factors of atherosclerosis, a history of smoking, diabetes, hypertension, and abnormal lipid profile have been shown to be important (7). In patients with juvenile SLE, smoking, diabetes, and uncontrolled hypertension are not common and therefore abnormal lipid profiles may be the most important risk factor.The lipid profile of both children and adults with SLE is the result of a combination of the influences of active disease, therapies, and genetics. The best way to determine the maximal potential effect of disease activity itself would be to examine patients at the time of presentation of SLE, when they are likely to have high disease activity but no effect of corticosteroid therapy.Studies in patients with active SLE suggested that there is a distinct pattern of lipid abnormalities of increased very low-density lipoprotein (VLDL) and triglycerides and decreased high-density lipoprotein (HDL-C), cholesterol and apolipoprotein A1 levels ("active SLE pattern")

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are diagnosed according to 2019 European League against Rheumatism (EULAR) /American College of Rheumatology (ACR) SLE classification criteria .
2. Patients diagnosed with jSLE between 5 and 18 years of age

Exclusion Criteria:

* 1. Patients on lipid lowering drugs for any other reason. 2. Patients with other autoimmune disease.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: .Patients diagnosed with jSLE between 5 and 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
lipid profile | 2 years
  pattern and frequency of dyslipoproteinemia in patients with newly diagnosed JSLE .
lipid profile | 2 years
  effect of disease activity on lipid profile of patients with JSLE

CONTACTS AND LOCATIONS:
Overall Officials: Jaafar I Mohamad, professor, Principal Investigator — Assiut University; Naglaa S Mohamad, lecturer, Principal Investigator — Assiut University; Yosra M Mamdouh, lecturer, Principal Investigator — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Sarkissian T, Beyene J, Feldman B, McCrindle B, Silverman ED. Longitudinal examination of lipid profiles in pediatric systemic lupus erythematosus. Arthritis Rheum. 2007 Feb;56(2):631-8. doi: 10.1002/art.22332. PMID 17265498
- [Background] Tyrrell PN, Beyene J, Benseler SM, Sarkissian T, Silverman ED. Predictors of lipid abnormalities in children with new-onset systemic lupus erythematosus. J Rheumatol. 2007 Oct;34(10):2112-9. Epub 2007 Sep 1. PMID 17787042
- [Background] Machado D, Sarni RO, Abad TT, Silva SG, Khazaal EJ, Hix S, Correia MS, Suano-Souza FI, Len CA, Terreri MT. Lipid profile among girls with systemic lupus erythematosus. Rheumatol Int. 2017 Jan;37(1):43-48. doi: 10.1007/s00296-015-3393-z. Epub 2015 Nov 16. PMID 26573664
- [Background] Rodrigues WDR, Sarni ROS, Abad TTO, Silva SGLD, Souza FIS, Len CA, Terreri MT. Lipid profile of pediatric patients with chronic rheumatic diseases - a retrospective analysis. Rev Assoc Med Bras (1992). 2020 Aug;66(8):1093-1099. doi: 10.1590/1806-9282.66.8.1093. PMID 32935804
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/17265498/